CLINICAL TRIAL: NCT03057574
Title: An Interventional Study to Assess the Efficacy and Safety of Gonapure® in Multifollicular Stimulation in Egyptian Women Undergoing IVF/ICSI
Brief Title: Gonapure® in Multifollicular Stimulation in Egyptian Women Undergoing IVF/ICSI
Acronym: GIVF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MinaPharm Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: r-hFSH13082013
Record Dates: First submitted 2016-11-30; First posted 2017-02-20 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female | interventions — follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Follitropin Alfa (Gonapure)
  Interventions: Drug: Follitropin Alfa

INTERVENTIONS:
Drug: Follitropin Alfa — Patients must be prescribed Follitropin Alfa (Gonapure®)
  Other Names: Gonapure ®

SUMMARY:
This study aims to record Efficacy, Safety and tolerability of Gonapure® prescribed for female subjects with infertility Undergoing IVF/ICSI

DETAILED DESCRIPTION:
Gonapure® is a human follicle stimulating hormone (FSH) preparation of recombinant DNA origin and contains no luteinizing hormone (LH) activity.

FSH stimulates ovarian follicular growth in women who do not have primary ovarian failure. FSH, the active component of Gonapure® is the primary hormone responsible for follicular recruitment and development. In order to affect final maturation of the follicle and ovulation in the absence of an endogenous LH surge, human chorionic gonadotropin (hCG) must be given following the administration of FSH, when monitoring of the patient indicates that sufficient follicular development has occurred. There is inter-patient variability in response to FSH administration.

The dosage and schedule of treatment for female infertility must be determined according to the needs of each patient; it is usual to monitor response by studying the patient's serum oestrogen level and/or by ultrasonic visualization of follicles.

Treatment should be started within the first 7 days of the menstrual cycle. Treatment is usually begun with 75 to 450 International units daily by intramuscular injection for 7 to 10 days; followed by individual adjustments according to the patient's follicular response i.e. until an adequate, but not excessive, response is achieved.

The investigator will decide the starting dose according to the standard clinical practice (and within the approved label).

Treatment is then stopped and followed after 1 or 2 days by a single dose of human chorionic Gonadotropin 10000 International units to induce oocyte maturation.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects aged between 18 and 38 years.
2. Female subjects with body mass index (BMI) ≥ 18 and ≤ 40 kilogram per square meter (kg/m^2)
3. Female subjects with basal FSH less than 10 IU/L and PRL serum values within the normal range in the early follicular phase.
4. Female subjects having both ovaries.
5. Female subjects with normal uterine cavity, which in the investigator's opinion is compatible with pregnancy.
6. Female subjects who have at least 1 wash-out cycle (defined as greater than or equal to 30 days since the last dose of clomiphene citrate or gonadotrophin treatment) since the last ART cycle and/or clomiphene citrate or gonadotrophin treatment prior to starting gonadotropin releasing hormone (GnRH) agonist therapy.
7. Female subjects who are willing and able to comply with the protocol for the duration of the trial
8. Female subjects who have given written informed consent, prior to any trial-related procedure, with the understanding that consent may be withdrawn by the subject at any time without prejudice to her future medical care.

Exclusion Criteria:

1. Female subjects with any medical condition, which in the judgment of the investigator may interfere with the absorption, distribution, metabolism or excretion of the drug.
2. Female subjects with uterine myoma requiring treatment.
3. Female subjects with any contraindication of being pregnant and/or carrying a pregnancy to term.
4. Female subjects with history of tumors of the hypothalamus and pituitary gland.
5. Female subjects with history of ovarian, uterine or mammary cancer.
6. Female subjects with history of hypersensitivity to the active substance follitropin alpha, FSH, or to any of the excipients of Gonapure ®.
7. Female subjects with untreated hydrosalpinx diagnosed by U/S.
8. Female subjects with abnormal gynecological bleeding of unknown etiology.
9. Female subjects with any medical condition which, in the opinion of the investigator, would prevent an effective response, such as primary ovarian failure, or malformations of the reproductive organs incompatible with pregnancy.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes retrieved on the day of Ovum Pick-Up | 50 days after baseline visit (EOS)
Number of Mature Oocytes (MII) Retrieved Per Participant | 50 days after baseline visit (EOS)
  Metaphase II (MII): The oocyte is in the second phase of meiosis and is mature. Oocytes at this stage of maturity are ready for fertilization.
  Mean number of Mature oocytes (MII) retrieved on the day of ovum pick up (OPU) will be calculated. Oocyte retrieval is a technique used in in-vitro fertilization in order to remove oocytes from the ovary of the female, enabling fertilization outside the body.
Quality of Oocytes Retrieved per participant | 50 days after baseline visit (EOS)
  It is graded on a good-fair-poor scale:
  * Good
    * Clear cytoplasm/normal shape
    * Single distinct polar body
    * Clear/thin zona pellucida
  * Fair
  * Slightly grainy cytoplasm/misshapen
  * Fragmented/abnormal polar body
  * Slightly pigmented/amorphous zona
  * Cytoplasmic bodies
  * PV (vitelline platelets) debris
  * Poor
    * Dark/grainy cytoplasm/misshapen
    * >1 polar body structure
    * Pigmented/thickened zona
    * Vacuoles
    * PV (vitelline platelets) debris
  * Good Quality embryos per participant. Those embryos that have reached the most advanced developmental stage and have the least cellular fragmentation (Grades "A" and/or "B") will be considered Good Quality embryos and will be selected for transfer.
  * Number of transferred embryos per participant.
  * Percentage of Participants with Clinical Pregnancy. Clinical pregnancy is defined by the number of sacs and hearts with activity per ultrasound scan.

SECONDARY OUTCOMES:
Eventual AE/SAEs related to the administration of Gonapure® | 50 days after baseline visit (EOS)
Total & Mean Gonapure ® Daily Dose | 14 days
  Time Frame: Start of treatment until end of stimulation cycle
Number of follicles ≥ 18 mm on day of administration of hCG | 50 days after baseline visit (EOS)
Number of Participants with Multiple Pregnancies | 50 days after baseline visit (EOS)
  Multiple pregnancies were defined as 2 or more fetal hearts with activity.
Number of Participants with Ovarian Hyperstimulation Syndrome | 50 days after baseline visit (EOS)
  OHSS is a syndrome which can manifest with enlarged ovaries, advanced ascites with increased vascular permeability, pleural fluid Accumulation, hemoconcentration, and increased blood clotting.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Kortam, PhD, Principal Investigator — Ain Shams University
Locations (2):
- Egypt (2):
  - Alexandria University, Alexandria
  - Ain Shams University, Cairo

IPD SHARING:
Plan to Share IPD: No